CLINICAL TRIAL: NCT03342924
Title: Associations of Cognition, Fitness, and Body Composition Among Ethnic Minority Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: University of Tennessee (Other)
Responsible Party: Principal Investigator, Arlette Perry, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20120584
Record Dates: First submitted 2017-07-13; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Physical Activity; Cognitive Function 1, Social
Keywords: cognitive control; physical fitness; minority
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flanker test and physical fitness test (Experimental): Participants performed a computer-based Flanker Task measuring cognitive control and physical fitness tests: two-minute walk, vertical jump, one-minute curl-ups, and handgrip strength. Body composition variables included: body mass index, percent body fat, waist circumference, and sagittal abdominal height. General linear models were performed to evaluate impacts of physical fitness and body composition on cognition, adjusting for age and sex.
  Interventions: Other: Flanker Test and physical fitness test

INTERVENTIONS:
Other: Flanker Test and physical fitness test — Socioeconomic status was determined using a trichotomous index. Inbody was used to assess body composition. To assess physical fitness, certain field tests were implemented using devices to quantify precise actions of physicality. Cognitive control was assessed using a computer-based Flanker Task.

SUMMARY:
Cognitive Control is crucial for learning and development. This study examined the associations between cognitive control and physical fitness and body composition among ethnic minority children.

DETAILED DESCRIPTION:
Cognitive control, or executive function, refers to a subset of goal-directed processes that are involved in perception, memory, attention, behavioral inhibition, verbal reasoning, and monitoring of actions. These aspects of cognitive control have been shown to have a direct association with academic performance, particularly mathematics and literacy. Many social and environmental factors impact the maturation of cognitive control, which can affect the growth and behavioral development of children. Physical activity has been shown to improve the functioning of the prefrontal cortex, which plays a central role in cognitive functioning. Studies have shown that children have better cognitive skills and grades when given a regimen of regular physical activity as well as executive control. Aerobic fitness has been correlated with faster reaction times as well as more accurate responses and higher prefrontal brain activity, which can enhance visuomotor function and proactive inhibition. In addition to positive health benefits, physical fitness, a product of the regular physical activity, is found to be positively associated with self-esteem, academic performance, and cognitive control. Growing evidence suggests that cognitive control may be inversely associated with obesity in childhood, adulthood, and in the elderly. The current rate of childhood obesity in the U.S. is 31.8% with poor physical fitness levels and increased sedentary behaviors as major contributors to the problem. Pediatric obesity may have negative implications on cognition, specifically memory, psychomotor speed, reaction time, complex attention, executive function and cognitive flexibility with a potential for decreased awareness or motivation in girls specifically. Overweight, inactive children, when compared to normal weight, active children, have exhibited lower planning and attention scores with detrimental effects on inhibitory control and psychosocial outcomes among girls ages nine to fifteen While new information continues to support the negative association between obesity and cognitive function, the direction of the relationship remains unclear. The extant literature also suggests that there is an inverse relationship between socioeconomic status and obesity and cognition. A recent study supported the influence of BMI on child executive control and BMI's inverse correlation with income, academic readiness, social competence and behavioral adjustment. Another study showed that white non-Hispanic and Hispanic children in fifth and seventh grades with lower socioeconomic status had a higher rate of obesity with inverse relationship most apparent in White non-Hispanic girls and fifth-grade Hispanic boys. A negative association has been observed between obesity and pattern construction in boys and vocabulary and pattern construction in girls. While there have been cross-sectional and randomized clinical trial studies correlating obesity and fitness with cognitive control, these studies fail to evaluate diverse racial/ethnic minority populations. Incorporating minority groups and gender differences into these associations are very important in generalizing findings to diverse demographics. Given the paucity of research examining the cumulative impact of obesity and physical fitness on cognition among diverse children, this study seeks to address gaps in the literature. This study utilized a comprehensive field test battery to evaluate associations among body composition, cardiovascular endurance, muscular strength and endurance, and motor skills, on executive control with gender, age, and race/ethnicity as mediators. This study is particularly relevant for Hispanic and African-American youth who show high rates of overweight and obesity

ELIGIBILITY:
Inclusion Criteria:

* Children were included in the study if they were: eight to 12 years old, and ethnic minority (Black and/or Hispanic/Latino), enrolled in YMCA after-school programs, able to engage in physical activities, had normal (or corrected to normal) vision based on the minimal 20/20 standard. Also, only children who were determined to be at Tanner Stages 1 or 2 (preadolescence) were included to account for the impact of puberty on measures of physical fitness and cognition.

Exclusion Criteria:

* Children who had prior or current metabolic, cardiovascular, or neurological disorders, and/or medication regimens that could interfere with evaluation of cognitive function were excluded from the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cognition | 8 weeks
  Cognitive control was assessed using a computer-based Flanker Task.

SECONDARY OUTCOMES:
Socioeconomic Status | 8 weeks
  Socioeconomic status was determined using a trichotomous index developed by Birnbaum et al. 2002 based on participation in free or reduced-price lunch program at school, the highest level of education attained by the mother and father, and the number of parents who worked full-time.
Aerobic Endurance | 8 weeks
  To assess physical fitness, certain field tests were implemented using devices to quantify precise actions of physicality. The NIH Toolbox two-minute Walk Endurance test was used to assess aerobic endurance.
Arm Strength | 8 weeks
  To assess physical fitness, certain field tests were implemented using devices to quantify precise actions of physicality.. A Jamar Plus handgrip dynamometer was used to assess right and left arm strength (kg).
Lower Body Power | 8 weeks
  To assess physical fitness, certain field tests were implemented using devices to quantify precise actions of physicality. To assess lower body power, a counter movement vertical jump was used.
Weight | 8 weeks
  The Inbody-520 multi-frequency bioimpedance analyzer was used to assess body composition. Information recorded included body weight, which was measured in pounds.
Waist Circumference | 8 weeks
  Waist circumference was used as a determinant of central obesity and was measured in centimeters using a Gulick spring loaded measuring tape.
Sagittal Abdominal Height | 8 weeks
  A portable anthropometer was used to measure sagittal abdominal height in centimeters as an indirect measure of visceral adiposity.
Percent Body Fat | 8 weeks
  The Inbody-520 multi-frequency bioimpedance analyzer was used to assess body composition. Information recorded included percent body fat.
Body Mass Index | 8 weeks
  The Inbody-520 multi-frequency bioimpedance analyzer was used to assess body composition. Information recorded included Body Mass Index.
Height | 8 weeks
  Height was measured using a Weigh Beam Eye-Level physicians' scale

CONTACTS AND LOCATIONS:
Overall Officials: Brian Anwari, Principal Investigator — University of Miami
Locations (1):
- Le Bonheur, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Only the study investigators and/or sponsor will monitor the plan for data and safety monitoring for this study. Shared data will be done through encrypted files and file management platform OneDrive.